CLINICAL TRIAL: NCT04782180
Title: Mobile Delivery of PrEP at a Syringe Services Program-A Pilot Study
Brief Title: PrEP at a Syringe Services Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Hansel Tookes, Professor of Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20210017
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hiv; Substance Use Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — emtricitabine tenofovir alafenamide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapid PrEP group (Experimental): Participants will receive PrEP i.e. Descovy for 12 months at the syringe services program.
  Interventions: Drug: Descovy 200Mg 25Mg Tablet; Behavioral: PrEP

INTERVENTIONS:
Drug: Descovy 200Mg 25Mg Tablet — daily Descovy tab by mouth
Behavioral: PrEP — PrEP will be provided in a community setting by community-based harm reduction program.

SUMMARY:
The purpose of this study is to see if providing participants with pre-exposure prophylaxis (PrEP) medicine right away at the IDEA Exchange will help participants remain in HIV negative.

ELIGIBILITY:
Inclusion Criteria:

1. over the age of 18
2. speak either English or Spanish
3. ability to provide informed consent
4. currently enrolled in the syringe services program
5. have a negative HIV rapid test result
6. estimated creatinine clearance > 30 ml/minute

Exclusion Criteria:

1. do not meet the above criteria of inclusion
2. decline to participate
3. test positive for HIV via rapid test
4. are pregnant or plan on becoming pregnant
5. have symptoms acute HIV.
6. Any other comorbidities that at the discretion of the investigator would prevent the participant from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self representation of gender identity
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hansel Tookes, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapid PrEP Group
Started | 90
Completed | 86
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rapid PrEP Group
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 4 participants consented and left before data was collected for baseline
  Participants
    number analyzed (Participants) | 86
    Female | 27
    Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 4 participants consented and left before data was collected for baseline
  Participants
    number analyzed (Participants) | 86
    Hispanic or Latino | 38
    Not Hispanic or Latino | 48
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 64
  More than one race | 7
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Intracellular Level of Tenofovir Diphosphate Levels Via Dried Blood Spot at 6-month Follow-up
Description: Tenofovir diphosphate levels will be quantified using a validated dried blood spot (DBS) assay. The outcome will be reported as the mean intracellular concentration (fmol/punch) at the 6-month follow-up visit. This measure reflects intracellular drug exposure and adherence.
Time Frame: 6 months
Population: Specimens were collected but none met laboratory acceptance criteria (insufficient punch volume and degradation). Therefore, no valid concentrations could be calculated. All values are reported as Not Analyzable.
Measure: Mean (Standard Deviation); unit: fmol/punch
Arm/Group | Rapid PrEP group
Number analyzed (Participants) | 86
fmol/punch | NA — No valid concentrations could be calculated because specimens failed laboratory acceptance criteria. Not applicable; no analyzable data are available

2. Secondary Outcome: Time to PrEP Initiation Post Negative HIV Rapid Test
Description: Number of days between receiving negative test result and initiating PrEP via self-report
Time Frame: up to 12 months
Population: All participants-initiated PrEP immediately following their negative test result. Because initiation occurred on the same day as the negative test (day 0), the calculated value for every participant was zero days
Measure: Number; unit: days
Arm/Group | Rapid PrEP group
Number analyzed (Participants) | 86
days | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rapid PrEP Group
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT04782180/Prot_SAP_000.pdf